CLINICAL TRIAL: NCT06350890
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Study Evaluating the Efficacy and Safety of HTD1801 in Patients With Type 2 Diabetes Mellitus Who Have Poor Glycemic Control After Dietary and Exercise Interventions
Brief Title: Efficacy and Safety of Berberine Ursodeoxycholate (HTD1801) in Patients With Type 2 Diabetes
Acronym: SYMPHONY-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HighTide Biopharma Pty Ltd (Industry)
Collaborators: Shenzhen HighTide Biopharmaceutical Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTD1801.PCT105
Record Dates: First submitted 2024-03-27; First posted 2024-04-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HTD1801 (Experimental): Administered orally twice daily (BID)
  Interventions: Drug: HTD1801
- Placebo (Placebo Comparator): Administered orally BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HTD1801 — HTD1801 1000 mg administered orally BID as four capsules
  Other Names: berberine ursodeoxycholate
  Arms: HTD1801
Drug: Placebo — Matching placebo administered orally BID as four capsules
  Arms: Placebo

SUMMARY:
The goal of this clinical study is to evaluate the efficacy and safety of Berberine Ursodeoxycholate (HTD1801) compared to placebo in patients with type 2 diabetes, inadequately controlled with diet and exercise alone.

DETAILED DESCRIPTION:
This Phase 3 randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of HTD1801 in two phases, a 24-week double-blind phase followed by a 28-week open-label extension. To ensure stabilization of glycemic control, eligible patients will first participate in a 4-week single-blind run-in period where investigators will provide guidance on lifestyle modification, concomitant medications, and procedures for self-monitoring of blood glucose. Following this period, patient eligibility will be reassessed. Eligible patients will then be randomized 2:1 to receive HTD1801 1000 mg twice daily (BID) or placebo for 24 weeks.

Patients who complete the double-blind treatment period will enter an open-label extension period where all patients will receive HTD1801 1000 mg BID for an additional 28 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Have been diagnosed with Type 2 diabetes mellitus
* Have followed dietary and exercise interventions for at least 8 weeks prior to screening
* If used any glucose-lowering drugs within the 8 weeks prior to screening such use was ≤7 days and was discontinued at least 4 weeks prior to screening
* Have HbA1c ≥7.5% to ≤11.0% (screening) and ≥7.0% to ≤10.5% (pre-randomization)
* Have fasting plasma glucose ≤13.9 mmol/L (screening and pre-randomization)
* Have a body mass index ≥19.0 kg/m^2 to ≤35.0 kg/m^2

Key Exclusion Criteria:

* Have type 1 diabetes
* Have had any acute diabetic complications within 12 months prior to screening
* Have had any Grade 3 hypoglycemic event within 12 months prior to screening
* Have had proliferative retinopathy or macular degeneration, severe diabetic neuropathy, or diabetic foot
* Have been taking any weight loss medication or dietary supplement, have participated in a weight loss program, or have adhered to a special diet within 12 weeks prior to screening
* Have used insulin or an insulin analogue for more than 14 days within 12 months prior to screening
* Have used any hypoglycemic drug during the 4-week run-in period prior to randomization
* Have had weight gain or loss ≥5% during the 4-week run-in period prior to randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: Mean Change in HbA1c | 24 Weeks
  Mean change in HbA1c from baseline to Week 24

SECONDARY OUTCOMES:
Double Blind (DB) Phase: Mean Change in Fasting Plasma Glucose | 24 Weeks
  Mean change in fasting plasma glucose from baseline to Week 24
DB Phase: Mean Change in 2-Hour Postprandial Glucose | 24 Weeks
  Mean change in 2-hour postprandial glucose from baseline to Week 24
DB Phase: Proportion of patients achieving HbA1c <7.0% | 24 Weeks
  Proportion of patients achieving HbA1c target values of <7.0% at Week 24
DB Phase: Proportion of patients achieving HbA1c <6.5% | 24 Weeks
  Proportion of patients achieving HbA1c target values of <6.5% at Week 24
DB Phase: Mean Change in Insulin Sensitivity (HOMA-IR) | 24 Weeks
  Mean change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) from baseline to Week 24
DB Phase: Mean Change in Low-Density Lipoprotein Cholesterol (LDL-C) | 24 Weeks
  Mean change in LDL-C from baseline to Week 24

OTHER OUTCOMES:
Open Label Extension (OLE) Phase: Mean Change in HbA1c | 52 weeks
  Mean change in HbA1c from baseline to Week 52
OLE Phase: Mean change in 2-Hour Postprandial Glucose | 52 Weeks
  Mean change in 2-hour postprandial glucose from baseline to Week 52
OLE Phase: Proportion of patients achieving HbA1c <7.0% | 52 Weeks
  Proportion of patients achieving HbA1c target values of <7.0% at Week 52
OLE Phase: Proportion of patients achieving HbA1c <6.5% | 52 Weeks
  Proportion of patients achieving HbA1c target values of <6.5% at Week 52
OLE Phase: Mean Change in Insulin Sensitivity (HOMA-IR) | 52 Weeks
  Mean change in HOMA-IR from baseline to Week 52
OLE Phase: Mean Change in LDL-C | 52 Weeks
  Mean change in LDL-C from baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Kui Liu, MD, Study Director — Shenzhen HighTide Biopharmaceutical Ltd.
Locations (56):
- China (56):
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - Beijing Pinggu Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital, CAMS & PUMC, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Handan First Hospital, Handan, Hebei
  - Hengshui People's Hospital (Harrison International Peace Hospital), Hengshui, Hebei
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Hospital of Qiqihar, Qiqihar, Heilongjiang
  - The Third Affiliated Hospital of Qiqihar Medical University, Qiqihar, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science & Technology (Jinghua), Luoyang, Henan
  - The First Affiliated Hospital of Henan University of Science & Technology (Kaiyuan), Luoyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - Zhumadian Central Hospital, Zhumadian, Henan
  - Huangshi Central Hospital, Huangshi, Hubei
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - The First People's Hospital of Changde City, Changde, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Yueyang People's Hospital, Yueyang, Hunan
  - Baotou City Central Hospital, Baotou, Inner Mongolia
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Nanjing Drum Tower Hospital - The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Sir Run Run Shaw Hospital Nanjing Medical University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Tonghua Central Hospital, Tonghua, Jilin
  - Panjin Liaohe Oilfield Gem Flower Hospital, Panjin, Liaoning
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - Qinghai Provincial People's Hospital, Xining, Qinghai
  - The Second Affiliated Hospital of Shaanxi University of Chinese Medicine, Xianyang, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Shanghai East Hospital of Tongji University, Shanghai, Shanghai Municipality
  - The Third People's Hospital of Datong, Datong, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - People's Hospital of Tianjin, Tianjin, Tianjin Municipality
  - The First People's Hospital of Kashi, Kashgar, Xinjiang
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Huzhou Central Hospital, Huzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No